CLINICAL TRIAL: NCT05869994
Title: Evaluation of Autologous Natural Killer Cell Activity in Primary Cancer Cell Cultures
Status: Withdrawn | Type: Observational
Why Stopped: Inactive study
Sponsor: Sarcoma Oncology Research Center, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: SOC-2205
Record Dates: First submitted 2023-01-20; First posted 2023-05-23 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor specimens from patients with sarcoma who are scheduled for elective surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of the study is to evaluate the anti-tumor activity of autologous natural killer cells in cultures of cancer cells obtained from patient's own tumor.

DETAILED DESCRIPTION:
The objectives of the study is to evaluate the anti-tumor activity of autologous natural killer cells in cultures of cancer cells obtained from patient's own tumor.

Study Design:

One hundred mL of blood will be collected in an EDTA container and transported to the laboratory for in vitro isolation and expansion of NK cell cultures.

Two or three weeks later, 25 cu mm of the patient's own tumor will be collected in PBS and transported to the laboratory for co-culture with autologous expanded and enhanced NK cells.

Inclusion Criteria:

Individuals must meet all of the inclusion criteria in order to be eligible to participate in the study, as follows:

* Male or Female ≥ 18 years of age
* Pathologically confirmed diagnosis of locally advanced unresectable or metastatic soft tissue sarcoma
* Patients who are already scheduled for surgery
* Ability to understand the purposes and risks of the study and has signed and dated a written informed consent form approved by the investigator's IRB/Ethics Committee
* Willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria: Patients who do not meet the inclusion criteria.

Methodology:

Male and female subjects > 18 years of age, of any ethnicity, with advanced soft tissue sarcoma will be recruited via patient referrals from the medical community, patient request for participation through internet research, patients being treated at the Sarcoma Oncology Research.

Study Duration:

The study is expected to take 24-30 months

Statistical Analysis Plan For the in vitro studies, multiple group comparisons at a single time point will be made via the independent analysis of variance (ANOVA) test, followed by Tukey's HSD test as a post-hoc test where appropriate. Assuming the required statistical power of 0.9 with a significance level of 0.05 and effect size of 0.4, an equal sample size of at least 19 is suggested for each group: 1) Untreated, 2) CH-SCP, 3) Nk cells and 4) CH-SCP-NK-based hydrogel. Differences in mean tumor growth and survival rate between the control and experimental groups at each time point will be tested with independent ANOVA followed by Tukey's HSD test as a post-hoc analysis where appropriate.

Baseline Descriptive Statistics Demographics, age, ethnicity, subtypes of sarcoma, number of patients, patients with locally advanced or metastatic will be described using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the inclusion criteria in order to be eligible to participate in the study, as follows:

  * Male or Female ≥ 18 years of age
  * Pathologically confirmed diagnosis of locally advanced unresectable or metastatic soft tissue sarcoma
  * Patients who are already scheduled for surgery
  * Ability to understand the purposes and risks of the study and has signed and dated a written informed consent form approved by the investigator's IRB/Ethics Committee
  * Willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

Patients who do not meet inclusion criteria.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female subjects > 18 years of age, of any ethnicity, with advanced soft tissue sarcoma will be recruited via patient referrals from the medical community, patient request for participation through internet research, patients being treated at the Sarcoma Oncology Research.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Antitumor activity | 1 month
  Inhibition of autologous cancer cell growth in vitro by autologous natural killer cells using an automated cell counter. For the in vitro studies, multiple group comparisons at a single time point will be made via the independent analysis of variance (ANOVA) test, followed by Tukey's HSD test as a post-hoc test where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Erlinda M Gordon, MD, Principal Investigator — Sarcoma Oncology Research Center
Locations (1):
- Sarcoma Oncology Research Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monette A, Ceccaldi C, Assaad E, Lerouge S, Lapointe R. Chitosan thermogels for local expansion and delivery of tumor-specific T lymphocytes towards enhanced cancer immunotherapies. Biomaterials. 2016 Jan;75:237-249. doi: 10.1016/j.biomaterials.2015.10.021. Epub 2015 Oct 9. PMID 26513416